CLINICAL TRIAL: NCT02396264
Title: Mediterranean Diet: A New Nutritional Approach for the Treatment of Normal Weight Women With Polycystic Ovary Syndrome (PCOS)?
Brief Title: Mediterranean Diet as Treatment for Normal Weight Women With PCOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona (Other)
Collaborators: Federico II University (Other); University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Francesco Orio, prof, Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIEMED2
Record Dates: First submitted 2015-03-08; First posted 2015-03-24 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Mediterranean Diet; Ovarian Cysts; Treatment; Ovarian Diseases; normocaloric diet
MeSH Terms: conditions — Polycystic Ovary Syndrome; Ovarian Cysts; Ovarian Diseases | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mediterranean Diet (Experimental): The diet programme will be characterized by carbohydrates (60 %); proteins (20 %, half comprised of vegetable proteins); total fat (20 %; saturated fat < 10 %). After calculating the patient's energy need, the amount of calories will be successively adjusted to mantain the same weight of the time of recruitment
  Interventions: Other: mediterranean diet
- normocaloric diet (Active Comparator): 50% carbohydrates, 30% total lipids and 20% proteins. After calculating the patient's energy need, the amount of calories will be successively adjusted to mantain the same weight of the time of recruitment
  Interventions: Other: normocaloric diet

INTERVENTIONS:
Other: mediterranean diet — 50 pcos women will be assigned to normocaloric mediterranean diet for 6 months
  Arms: Mediterranean Diet
Other: normocaloric diet — 50 pcos women will be assigned to standardized normocaloric diet for 6 months
  Arms: normocaloric diet

SUMMARY:
Polycystic ovary syndrome (PCOS) is the most common endocrinopathy of reproductive-aged women characterized by chronic anovulation, hyperandrogenism and insulin resistance. Available guidelines recommend lifestyle intervention although they do not suggest the best dietetic regimen for the treatment of PCOS. Thus, the purpose of this study is to compare the effectiveness of two nutritional protocols, namely Mediterranean Diet and standardized normocaloric Diet in normal weight women with PCOS.

DETAILED DESCRIPTION:
PCOS is the most common endocrine disorder of reproductive age women, that is often characterized by chronic anovulation, hyperandrogenism and insulin resistance. The central importance of insulin resistance in the pathogenesis of the syndrome has been established by several in vivo and in vitro studies. No data are available for the best therapeutical approach for metabolic dysfunction of PCOS. In addition, although insulin resistance is a crucial pathogenetic factor for PCOS and lifestyle change program improves insulin resistance, no available data can also suggest whether non-obese women with PCOS benefit or did not from lifestyle change program including diet without calorie-restriction. Although there are not studies focused on the effectiveness and safety of Mediterranean diet in PCOS, several indirect studies performed in obese and/or insulin resistant subjects, seem to suggest a potential role of this diet in PCOS population and, in particular, on long-term PCOS-related health risk. In this study, the investigators' purpose is to compare two nutritional protocols in order to find the best dietetic approach for improving clinical, metabolic and hormonal outcomes in normal weight women with PCOS.

ELIGIBILITY:
Inclusion Criteria: Polycystic ovary syndrome (using ESHRE/ARSM 2007 criteria), 18 ≤BMI ≤ 25

Exclusion Criteria: Age <18 or >35 years, BMI less than 18 and higher than 25, Pregnancy, Hypothyroidism, hyperprolactinemia, Cushing's syndrome, nonclassical congenital adrenal hyperplasia, use of oral contraceptives, glucocorticoids, antiandrogens, ovulation induction agents, antidiabetic or antiobesity drugs or other hormonal drugs within the previous 6 months, neoplastic, metabolic (including glucose intolerance), hepatic, and cardiovascular disorder or other concurrent medical illness (i.e. diabetes, renal disease, or malabsorptive disorders, cephalea).

-

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
improvement in insulin resistance measured by HOMA index | 6 months

SECONDARY OUTCOMES:
improvement in clinical parameters (Body mass index, normalization of menses, hirsutism, waist to hip ratio) | 6 months
improvement in metabolic parameters(total, LDL and HDL cholesterol) | 6 months
improvment in hormonal parameters (Testosterone, Androstenedione, DHEAS, FSH, LH, beta estradiol) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Orio, MD, Principal Investigator — Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona
Locations (1):
- Fertility Techniques SSD,Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona, Salerno, Salerno, Italy

REFERENCES:
- [Result] Orio F, Palomba S. Reproductive endocrinology: New guidelines for the diagnosis and treatment of PCOS. Nat Rev Endocrinol. 2014 Mar;10(3):130-2. doi: 10.1038/nrendo.2013.248. Epub 2013 Dec 10. PMID 24322653
- [Result] Boghossian NS, Yeung EH, Mumford SL, Zhang C, Gaskins AJ, Wactawski-Wende J, Schisterman EF; BioCycle Study Group. Adherence to the Mediterranean diet and body fat distribution in reproductive aged women. Eur J Clin Nutr. 2013 Mar;67(3):289-94. doi: 10.1038/ejcn.2013.4. Epub 2013 Feb 6. PMID 23388669
- [Result] Abiemo EE, Alonso A, Nettleton JA, Steffen LM, Bertoni AG, Jain A, Lutsey PL. Relationships of the Mediterranean dietary pattern with insulin resistance and diabetes incidence in the Multi-Ethnic Study of Atherosclerosis (MESA). Br J Nutr. 2013 Apr 28;109(8):1490-7. doi: 10.1017/S0007114512003339. Epub 2012 Aug 30. PMID 22932232
- [Derived] Hooper L, Abdelhamid AS, Jimoh OF, Bunn D, Skeaff CM. Effects of total fat intake on body fatness in adults. Cochrane Database Syst Rev. 2020 Jun 1;6(6):CD013636. doi: 10.1002/14651858.CD013636. PMID 32476140